CLINICAL TRIAL: NCT04019236
Title: Effect of Implementing Nursing Care on Breathing Discomfort and Its Outcomes Among Mechanically Ventilated Patients
Brief Title: Nursing Care for Breathing Discomfort Among Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Mamdouh Aziz soliman, Principal Investigator, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Dyspnea among MV Pts
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: Researcher will provide patients with suitable care for relieving dyspnea and record the outcomes
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- " interventional " (Other): New other than Routine nursing care will be used.
  Interventions: Other: visual analogue scale (VAS),Respiratory distress observational scale (RDOS) and other Nursing care
- " Control group " (No Intervention): Routine care only will be done for this group

INTERVENTIONS:
Other: visual analogue scale (VAS),Respiratory distress observational scale (RDOS) and other Nursing care — Distressed patient will be assessed by visual analogue scale(VAS) or respiratory distress observational scale.Nursing interventions will be done according to its causes as giving supplemental O2 therapy, pharmacologic therapy ,initiating positive pressure ventilation or change Ventilator settings (TV, PEEP, Inspiratory pressure ), Improve inspiratory muscle function by Nutrition, positioning or by minimizing use of steroids , clearing airway by Suctioning, Check O2 saturation level frequently and maintain O2 saturation between 95-100%, ,Raising the HOB (Head of the Bed), high Fowler's ,Give pain medications as prescribed or diuretics as ordered and If thick secretions increase oral fluids intake
  Arms: " interventional "

SUMMARY:
Breathing discomfort (dyspnea) during mechanical ventilation in the ICU may complicate care.

DETAILED DESCRIPTION:
Patients on ventilators experience a variety of discomforts: symptoms (dyspnea ,fatigue , pain ) ,emotions (depression, anxiety ,panic) and feeling of lack to control .Patients may or may not express this discomfort outwardly with agitation ,restlessness ,grimacing or increase in the vital signs (heart rate ,blood pressure ,breathing frequency).The aim of the present study is to assess the prevalence of dyspnea among mechanically ventilated patients, Describe interventions that may alleviate breathing discomfort and examine its impact on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Intubated or tracheostomized patients who were mechanically ventilated for >24 hrs.
* Age : 18-60 yrs
* Patients with Respiratory diseases
* Patients during spontaneous breathing trial

Exclusion Criteria:

* • Patients with acidosis, anemia ,drug poisoning,psychogenic disorders or neuro-muscular disorders

  * (non invasive ventilation)NIV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of breathing discomfort among Mechanically ventilated patients | 1year
  visual analogue scale "VAS" for conscious patients and respiratory observational distress scale "RDOS" for unconscious patients
Effect of nursing intervention on patient and ICU | 1year
  Clinical outcomes "length of stay,type of discharge or other morbidities"

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of nursing, Asyut, Egypt

REFERENCES:
- [Background] Persichini R, Gay F, Schmidt M, Mayaux J, Demoule A, Morelot-Panzini C, Similowski T. Diagnostic Accuracy of Respiratory Distress Observation Scales as Surrogates of Dyspnea Self-report in Intensive Care Unit Patients. Anesthesiology. 2015 Oct;123(4):830-7. doi: 10.1097/ALN.0000000000000805. PMID 26259140
- [Background] Zhuang Q, Yang GM, Neo SH, Cheung YB. Validity, Reliability, and Diagnostic Accuracy of the Respiratory Distress Observation Scale for Assessment of Dyspnea in Adult Palliative Care Patients. J Pain Symptom Manage. 2019 Feb;57(2):304-310. doi: 10.1016/j.jpainsymman.2018.10.506. Epub 2018 Nov 2. PMID 30391404
- [Background] Puntillo K, Nelson JE, Weissman D, Curtis R, Weiss S, Frontera J, Gabriel M, Hays R, Lustbader D, Mosenthal A, Mulkerin C, Ray D, Bassett R, Boss R, Brasel K, Campbell M. Palliative care in the ICU: relief of pain, dyspnea, and thirst--a report from the IPAL-ICU Advisory Board. Intensive Care Med. 2014 Feb;40(2):235-248. doi: 10.1007/s00134-013-3153-z. Epub 2013 Nov 26. PMID 24275901
- [Background] Campbell ML. Dyspnea. Crit Care Nurs Clin North Am. 2017 Dec;29(4):461-470. doi: 10.1016/j.cnc.2017.08.006. Epub 2017 Sep 23. PMID 29107308